CLINICAL TRIAL: NCT06690723
Title: Exploring the Synergistic Effect of Vitamin D and SGLT-2 Inhibitor on Cardio-metabolic Markers and the Renin Angiotensin Aldosterone System in CPAP-naive Obstructive Sleep Apnea Population
Brief Title: Vitamin D and SGLT-2 Inhibitor in CPAP-naive Obstructive Sleep Apnea
Acronym: D3DOSA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Malaysia Sarawak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNIMAS_OSA; FRGS/1/2021/SKK01/UNIMAS/02/1 (Other Grant/Funding Number: Ministry of Higher Education Malaysia FRGS); F05/IMPACT/2122/2021 (Other Grant/Funding Number: UNIMAS)
Record Dates: First submitted 2024-10-10; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive sleep apnea; Hypertension; Vitamin D; Sodium glucose transporter-2 inhibitor; Dapagliflozin; Endothelial function; Metabolic dysfunction associated steatotic liver disease; MASLD; Heart rate variability; Cardiac autonomic function
MeSH Terms: conditions — Sleep Apnea, Obstructive; Hypertension | interventions — dapagliflozin; Sodium-Glucose Transporter 2 Inhibitors; Cholecalciferol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Lifestyle modification (Active Comparator): Participants are taught about lifestyle modification including diet and exercise
  Interventions: Behavioral: Lifestyle modification
- Vitamin D3 (Cholecalciferol) (Active Comparator): Participants are given vitamin D3 for 16 weeks on top of lifestyle modification advice
  Interventions: Drug: Vitamin D3 ( Colecalciferol)
- Dapagliflozin (Forxiga) (Active Comparator): Participants are given Dapagliflozin 10mg daily for 16 weeks on top of lifestyle modification advice
  Interventions: Drug: Dapagliflozin (Forxiga)
- Vitamin D3 plus Dapagliflozin (Active Comparator): Participants are given vitamin D3 plus Dapagliflozin 10mg daily for 16 weeks on top of lifestyle modification advice
  Interventions: Drug: Vitamin D3 plus Dapagliflozin

INTERVENTIONS:
Drug: Dapagliflozin (Forxiga) — Dapagliflozin plus lifestyle modification
  Other Names: SGLT-2 inhibitor
  Arms: Dapagliflozin (Forxiga)
Drug: Vitamin D3 ( Colecalciferol) — Vitamin D3 plus lifestyle modification
  Arms: Vitamin D3 (Cholecalciferol)
Drug: Vitamin D3 plus Dapagliflozin — Vitamin D3 plus Dapagliflozin plus lifestyle modification
  Arms: Vitamin D3 plus Dapagliflozin
Behavioral: Lifestyle modification — Lifestyle modification alone
  Arms: Lifestyle modification

SUMMARY:
The purpose of this study is to determine if vitamin D supplement and SGLT-2 inhibitor treatment combination can improve cardiovascular risks in patients with OSA and hypertension, on top of lifestyle modification, before treatment with CPAP therapy.

It aims to answer if this treatment combination can improve i) renin-angiotensin-aldosterone system (RAAS) parameters, ii) cardio-metabolic risks iii) sleepiness symptoms and quality of life

Researchers will compare the outcome with 3 other groups of treatment: vitamin D supplementation and lifestyle modification, SGLT2-inhibitor and lifestyle modification, and lifestyle modification alone.

Participants will need to answer 2 questionnaires (Epworth Sleepiness Scale, WHO-quality of life), undergo anthropometric measurements (blood pressure, pulse rate, weight, height, waist circumference, neck circumference), blood taking (aldosterone, renin, vitamin D, calcium, albumin, phosphate, intact parathyroid hormone, kidney function, blood sugar, cholesterol and hsCRP), ultrasound of liver, ultrasound of blood vessel, and heart rate variability assessment using Polar H10 device and 24-hour Holter monitoring.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a medical condition that occurs in 25% to 58% of men and 10% to 37% of women. Close to 50% of express bus drivers in Malaysia were diagnosed with OSA. The association between obesity and OSA is compelling. Approximately 70% of individuals with OSA are obese; whereas prevalence of OSA in people with obesity is 40%. Every 10-kg body weight increment increases OSA risk twofold. As Malaysia has the highest prevalence of adult with obesity in South East Asia with 50% of our adult population being overweight or obese, this makes OSA a very common medical condition in our population. Among patients with obesity undergoing bariatric surgery in our local population, the prevalence of OSA was found to be 80.5%.

The link between renin-angiotensin-aldosterone system (RAAS) and OSA could be bi-directional. It is hypothesized that aldosterone causes salt and water retention leading to edema of the parapharyngeal tissues resulting in obstruction of upper airway and worsening of OSA symptoms. Recurring upper airway collapse in OSA also causes intermittent hypoxia, which increases plasma levels of both renin and aldosterone in animal models, and stimulation of the receptor in the carotid body in rats. The association between OSA and hyperaldosteronism is also believed to be contributed by other factors, including endothelial dysfunction and sympathetic nervous system (SNS) derangement.

Vitamin D plays an important role in calcium homeostasis and metabolism. It is involved in maintenance of calcium and phosphorus levels in the blood, and bone content. Vitamin D is also implicated in several non-skeletal conditions, such as cardiovascular disease, cancer, autoimmune disorders and diabetes mellitus. Vitamin D deficiency has been associated with worse cardiovascular outcomes. Hypovitaminosis D is related to increased risks of cardiovascular diseases, metabolic dysfunctions, and elevated all-cause mortality in the general population. Vitamin D deficiency augments RAAS leading to elevated aldosterone and lowered renin. This is supported by a reduction in aldosterone and an increase in plasma renin in patients with heart failure, arterial hypertension and primary aldosteronism when repleted with vitamin D.

Sleep fragmentation in patients with OSA due to nocturnal hypoxia can lead to daytime drowsiness and fatigue, causing a decrease in outdoor activities and, hence, a decrease in vitamin D synthesis. Moreover, repeated aggravation of upper airway obstruction and hypopnea in these patients partly inhibit vagal nerve activity, affect gastrointestinal motility and secretion of gastrointestinal hormones. These affect absorption and metabolism of vitamin D. Besides, sleep disturbances, intermittent hypoxia, upper airway obstruction and chronic increased abdominal pressure could result in gastroesophageal reflux and gastric ischemia, affecting vitamin D absorption.

Vitamin D receptor-knockout-mice demonstrated a marked increase in angiotensin II and renin levels, whereas 1-alpha-hydroxylase (enzyme needed to synthesize active vitamin D) deficiency enhanced RAAS activity, which was attenuated with administration of active vitamin D. Besides, vitamin D receptors have been found in adrenocortical tissues. Vitamin D3 is demonstrated to decrease expression and activity of the gene which encodes the enzyme required for aldosterone synthesis.

Sympathetic and parasympathetic nervous system interactively regulate visceral functions to maintain the body homeostatic milieu, and to enable reaction and adaptation to external and internal stressor stimuli.[63] Patients with OSA exhibit high levels of sympathetic activity during sleep as well as when awake. Aldosterone is found to augment sympathetic activity in patients with resistant hypertension.

Patients with OSA experience repetitive apneic events during sleep, with consequent hypoxia and hypercapnia. These act via chemoreflexes and baroreceptors to increase sympathetic activity. Night time chronic intermittent hypoxia also activates central nervous system and augments peripheral chemo-sensitivity, that are carried over into wakefulness, resulting in sustained daytime sympathetic over-activity. Heart rate variability (HRV) is a method that involves analysis of different parameters based on time variation between successive heart beats. HRV can be analyzed using time-domain analysis, based on the variations of cardiac cycles (RR interval) within a given time, and its parameters are obtained from statistical methods in the RR intervals such as mean, measures of dispersion, and count. In a healthy autonomic nervous system, there is a predominance of parasympathetic cardiac modulation at rest. Conversely, in individuals with heart disease, there is a greater sympathetic modulation and lesser parasympathetic modulation of the heart. HRV reflects the relationship between sympathetic and parasympathetic nervous system, which is a good predictor of future cardiovascular problems.

Endothelial dysfunction is a known risk factor for cardiovascular events. Vitamin D is known to have vaso-protective effect, while vitamin D deficiency leads to endothelial dysfunction. Vitamin D plays an essential role in endothelial function through 3 main pathways: i) regulate nitric oxide (NO) bioavailability, ii) anti-oxidant effect, and iii) anti-inflammatory effect. NO is a potent vasodilatory substance with important vaso-protective effect. Vitamin D reduces oxidative stress-induced endothelial dysfunction via regulating reactive oxygen species (ROS). Vitamin D deficiency leads to increased ROS production, which then inhibits NO synthesis, leading to endothelial dysfunction. Besides, vitamin D has an anti-inflammatory property and acts by suppressing pro-inflammatory markers to prevent endothelial dysfunction. Vitamin D also elicits anti-oxidant effects through upregulating expression of anti-oxidative enzymes.

Hypothesis The researchers postulate that, among patients with CPAP-naive obstructive sleep apnea (OSA) and hypertension, vitamin D supplement and SGLT2i treatment combination act as an effective adjunct treatment combination in

1. improving RAAS parameters
2. improving cardiometabolic indices
3. improving sleepiness symptoms and quality of life

Research objectives

1. To determine the role of vitamin D supplement and SGLT2i treatment combination in improving RAAS parameters among patients with obstructive sleep apnea (OSA) and hypertension
2. To ascertain the effect of vitamin D supplement and SGLT2i treatment combination on improving cardiometabolic indices among patients with CPAP-naive OSA
3. To evaluate the effect of vitamin D supplement and SGLT2i treatment combination on improving sleepiness symptoms and quality of life among patients with CPAP-naive OSA

I. Study Design Prospective, parallel, open-label, case-control II. Study Criteria INCLUSION CRITERIA

1. Aged 18 years and above
2. Consent to study
3. OSA confirmed on sleep study
4. Hypertension (SBP>140mmHg and/or DBP>90mmHg) or on anti-hypertensive EXCLUSION CRITERIA

1. Diagnosis of secondary hypertension 2. Undergone surgical or medical therapy for PA 3. Chronic kidney disease (eGFR<30ml/min/1.73m2) 4. Long term use of systemic steroids 5. Presence of thyroid dysfunction or suspected Cushing's syndrome 6. On current use of continuous positive airway pressure (CPAP) therapy for OSA 7. Recent myocardial infarction or stroke (within 6 weeks prior to study) 8. Congestive heart failure 9. Long-standing atrial fibrillation, ie atrial fibrillation >12 months in duration 10. On vitamin D supplements 11. On SGLT-2 inhibitor 12. Underlying type 1 diabetes or history of ketoacidosis 13. History of severe recurrent genito-urinary tract infections 14. History of, or increased risk of, bone fractures 15. Pregnant

III. Sample Size Sample size is calculated using G Power software. Assuming a moderate effect size (f=0.25) will be seen with the use vitamin D3 supplement and SGLT2i treatment combination, with 5% margin of error, 80% power, 124 participants with confirmed OSA and hypertension need to be recruited. Including estimated 20% of non-respondent rate, we aim to recruit 160 participants in total.

IV. Sampling Method (Consecutive Sampling) Ethical clearance will be obtained from Malaysia Medical Research and Ethics prior to conduct of study. All researchers will adhere to the Declaration of Helsinki and the Malaysian Good Clinical Practice Guidelines. Patients who are more than 18 years of age from the community, hospitals and clinics in Kuching, Samarahan and Serian will be invited to participate in this study if they fulfil the study criteria, after informed consent. The family medicine specialists of all clinics around Kuching and Samarahan will be informed about this study and patients who fulfil the study criteria will be referred to the research team. The clinics involved are Klinik Kesihatan Jalan Masjid, Batu Kawa, Sentosa, Petra Jaya, Samarahan and Tanah Puteh. The community will be reached out via research advertisement or poster on UNIMAS facebook page, or via community health screening. Patients who will be considered for recruitment include i) Those who are referred to the surgical clinic for bariatric surgery ii) Those who are referred to the Endocrine clinic for obesity iii) Those who are referred for suspected sleep apnea iv) Those who present to the health clinics or general medical clinic in Sarawak General Hospital for other medical conditions The research will be conducted in UNIMAS, Kota Samarahan and Sarawak General Hospital, Kuching.

Study participants will be approached by researchers to be recruited into the study. Informed consent will be obtained by principal investigator in research clinic of UNIMAS main campus. Study participants will be informed about i) Purpose of the study ii) Study procedure iii) Responsibilities of study participants iv) Risk and benefit v) Privacy and confidentiality vi) Voluntary participation Study participants will be given sufficient time to consider their participation in the study. The expected duration of participation for each study participant is 16 weeks.

The facilities available in the research sites include sleep laboratories, radiology unit, as well as endocrine, respiratory and cardiovascular clinics. Available expertise include endocrinologists, respiratory physicians, cardiologists, radiologists and medical scientist.

Anti-hypertensive will be switched to those with least effect on aldosterone and renin for at least 2 weeks before the start of research. Epworth Sleepiness Scale (ESS) will be documented at baseline. Their socio-demographic data will be collected and anthropometric measurements documented. If the participant has underlying hypertension, duration of hypertension and type of anti-hypertensive medications will be recorded. Seated clinic blood pressure will be measured using appropriately-sized cuff at each clinic visit after 5 minutes of rest. The mean of 2 readings will be recorded at visit 1 (V1).

Approximately 20ml of blood will be taken for aldosterone, renin, 25(OH)D, calcium, albumin, phosphate, intact parathyroid hormone (iPTH), renal profile, HbA1c, plasma glucose, lipid profile, and hsCRP at V1 and analyzed by a medical scientist. The results will be then interpreted by the principal investigator. Blood samples will not be used for pharmacogenomic analysis. Residual blood samples will be discarded together with the syringes and needles into the sharp bin. No blood specimens will be stored for future research.

Study participants will also fill in the World Health Organization abbreviated version of quality of life (WHOQOL-BREF) questionnaire to assess their quality of life with OSA. It consists of 26 items, covering four domains, ie physical health, psychological, social relationships, and environment. There are also two separate questions which ask specifically about the individual's overall perception of their health, and the individual's overall perception of their quality of life.

All study participants will undergo Polar H10 monitoring for assessment of short term HRV and subsequently have Holter monitor attached for 24 hours to assess long term HRV as indicators of cardiac autonomic function. HRV will be analyzed using time-domain analysis. The results will be analysed by a consultant cardiologist.

All study participants will also undergo ultrasound flow-mediated dilatation (FMD) of brachial artery to assess endothelial function, after a fast for at least 8 to 12 hours before the study, in a quiet, temperature-controlled room. All subjects should not exercise, should not ingest substances that might affect FMD such as caffeine, high-fat foods and vitamin D or use tobacco for at least 4 to 6 hours before the study. The subject will be positioned supine with the arm in a comfortable position for imaging the brachial artery. At the same setting, hepatobiliary ultrasound will be performed to detect presence of hepatic steatosis. This procedure will be performed and results analysed by a radiologist.

All study participants will be randomized via block randomization using computerized generation to receive lifestyle modification (Group 1, n=40) or lifestyle modification plus oral vitamin D supplement (Group 2, n=40) or lifestyle modification plus Dapagliflozin 10mg (Group 3, n=40) or lifestyle modification plus oral vitamin D3 plus Dapagliflozin 10mg (Group 4, n=40) for 16 weeks. Vitamin D deficiency is defined as serum 25(OH)D as <20ng/dL and vitamin D insufficiency is defined as serum 25(OH)D as <30ng/mL. In accordance with guideline, study participants with vitamin D deficiency or insufficiency will be given vitamin D3 6000IU a day then 4000IU/day if vitamin D level achieves 30ng/dL. Study participants who are vitamin D sufficient will be given vitamin D3 4000IU/day. Patient compliance of Vitamin D supplement will be monitored via pill counting during follow up visits. The risk for study participants is minimal. As inactivated vitamin D is given, calcium absorption can be regulated, hence the risk of excess calcium in blood is rare.

Study participants randomized to receive Dapagliflozin will be counseled on the possible side effects prior to initiation, ie increased urinary frequency, dehydration, genitourinary tract infection and rarely, ketoacidosis and bladder cancer. Participants will be advised to seek medical attention immediately if they develop features to suggest the above side effects. Dapagliflozin will be initiated at 10mg per day. For participants with underlying type 2 diabetes, dosage of other anti-diabetic treatment will be adjusted to reduce the risk of hypoglycemia with addition of Dapagliflozin. Throughout the study period, adjustment of other anti-diabetic treatment is allowed as per the managing clinicians' judgement. Patient compliance of Dapagliflozin will be monitored via pill counting during follow up visits.

Follow-up phone call will be made to study participants at 1-week and 4-week post treatment to inquire about tolerability to treatment and ensure compliance. Any adverse effects from the treatment will be documented during follow-up phone call and at every clinic visit.

Serum 25 (OH)D, calcium, albumin, phosphate, hsCRP, ultrasound FMD, ultrasound hepatobiliary system and Polar H10 monitoring will be repeated at 8 weeks. Vitamin D supplement dosage will be titrated if indicated. This is followed by anthropometric measurements and assessment (ESS, blood for aldosterone and renin, 25 (OH)D, calcium, albumin, phosphate, renal profile, plasma glucose, lipid profile, HbA1c, hsCRP, Polar H10, Holter, ultrasound FMD of brachial artery, hepatobiliary ultrasound and WHOQOL-BREF) at 16-week post-treatment.

No rescue medication or procedures are involved in this research.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years and above
2. Obstructive sleep apnea (OSA) confirmed on sleep study
3. Hypertension (SBP>140mmHg and/or DBP>90mmHg) or on anti-hypertensive

Exclusion Criteria:

1. Diagnosis of secondary hypertension
2. Undergone surgical or medical therapy for PA
3. Chronic kidney disease (eGFR<30ml/min/1.73m2)
4. Long term use of systemic steroids
5. Presence of thyroid dysfunction or suspected Cushing's syndrome
6. On current use of continuous positive airway pressure (CPAP) therapy for OSA
7. Recent myocardial infarction or stroke (within 6 weeks prior to study)
8. Congestive heart failure
9. Long-standing atrial fibrillation, ie atrial fibrillation >12 months in duration
10. On vitamin D supplements
11. On SGLT-2 inhibitor
12. Underlying type 1 diabetes or history of ketoacidosis
13. History of severe recurrent genito-urinary tract infections
14. History of, or increased risk of, bone fractures
15. Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2024-09-03 (Actual); Study Completion 2024-09-03 (Actual)

PRIMARY OUTCOMES:
hsCRP (mg/L) | 16 weeks
  To examine the effect of vitamin D supplement and SGLT2i treatment combination on improving hsCRP which reflect inflammation. The lower the hsCRP, the better the health outcomes
Endothelial function | 16 weeks
  To determine the effect of combining vitamin D3 and SGLT2i treatment combination in improving endothelial function assessed via ultrasound flow-mediated dilatation of brachial artery, where normal is >7.1%
Metabolic-associated steatotic liver disease | 16 weeks
  To evaluate the effect of vitamin D3 and SGLT2i treatment combination in improving steatotic liver disease, which are graded as normal, grade 1, grade 2, and grade 3
Heart rate variability | 16 weeks
  To evaluate the effect of vitamin D3 and SGLT2i treatment combination in improving heart rate variability (HRV) assessed via Polar H10 device (for short-term HRV) and 24-hour Holter monitoring (for long-term HRV).

SECONDARY OUTCOMES:
Plasma aldosterone levels (ng/dL) | 16 weeks
  To evaluate the role of vitamin D supplement and SGLT2i treatment combination in improving plasma aldosterone levels
Plasma renin levels (uIU/mL) | 16 weeks
  To determine the effect of vitamin D3 plus SGLT2i treatment combination in improving plasma renin levels
Sleepiness symptoms | 16 weeks
  To determine the role of vitamin D supplement and SGLT2i treatment combination in improving Epworth Sleepiness Score (minimum score 0, maximum score 24, the lower the score the better the outcome)
Quality of life | 16 weeks
  To determine the role of vitamin D supplement and SGLT2i treatment combination in improving World Health Organization quality of life scores (the higher the score, the better the quality of life)

CONTACTS AND LOCATIONS:
Locations (1):
- University Malaysia Sarawak, Sarawak, Sarawak, Malaysia

IPD SHARING:
Plan to Share IPD: No
Confidentiality

REFERENCES:
- [Derived] Loh HH, Tay SP, Koa AJ, Yong MC, Said A, Chai CS, Abdul Malik NM, Su AT, Tang BBC, Tan FHS, Sukor N. Unveiling the benefits of Vitamin D3 with SGLT-2 inhibitors for hypertensive obese obstructive sleep apnea patients. J Transl Med. 2025 Mar 7;23(1):296. doi: 10.1186/s12967-025-06312-w. PMID 40055713